CLINICAL TRIAL: NCT05474274
Title: Development of the PAIN (Pain AI iNtervention) Platform for Patients at Home
Brief Title: PAIN (Pain AI iNtervention) Platform for Patients at Home
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Other Study IDs: 21-013443
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pain
Keywords: Physiological markers for pain intensity; AI to objectively measure pain intensity; Medication over-use
MeSH Terms: conditions — Pain | interventions — Machine Learning Algorithms; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Surgery data collection system: Subjects undergoing standard of care low-risk plastic surgery be provided with wearable sensors to take home and start recording heart rate, body temperature and body movements
  Interventions: Other: Machine learning algorithms

INTERVENTIONS:
Other: Machine learning algorithms — Machine learning techniques to rank order physiologic variables obtained via the wearable and handheld devices as well as remove low-importance and redundant variables to accurately determine postoperative pain intensity in outpatients
  Other Names: Artificial Intelligence (AI) enabled system

SUMMARY:
The purpose of this research is to identify physiological markers to determine pain intensity and build an Artificial Intelligence (AI) enabled system to objectively measure pain intensity. Researchers hope to personalize pain medication regimens to help prevent medication over-use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing low-risk outpatient plastic surgery procedures with expected pain intensities ranging from mild to severe.

Exclusion Criteria:

* Patients with treated or untreated cardiopulmonary syndromes.
* Patients with treated or untreated ophthalmologic pathologies.
* Patients with skin pathologies that prevent us from using the TENS device.
* Patients with pathologies or conditions preventing them from appropriately using their voice.
* Patients with barriers to effective communication.
* Patients with poor digital literacy.
* Patients incapable of taking oral medication.
* Patients who are currently taking medical therapy for chronic pain.
* Patients with a previous diagnosis of severe anxiety disorders.
* Patients who are immobile at baseline.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older undergoing low-risk outpatient plastic surgery procedures with expected pain intensities ranging from mild to severe will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Using machine Learning for Postoperative Pain Pain Prediction | 8 months
  The primary outcome will be the accuracy of machine learning algorithms for postoperative pain prediction using root mean square errors.

SECONDARY OUTCOMES:
Physiologic variable %Δ defining the physiologic biomarker's change in measurements after pain medication | 8 months
  The secondary outcome will be the physiologic variable's use to define the physiologic biomarker's change in measurements after pain medication (%Δ in signal's respective units).
Physiologic variable absolute Δ defining the physiologic biomarker's change in measurements after pain medication | 8 months
  The secondary outcome will be the physiologic variable's use to define the physiologic biomarker's change in measurements after pain medication (absolute Δ in signal's respective units).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials